CLINICAL TRIAL: NCT05438745
Title: The Effects of Dog Therapy on Ambulance Staff Burnout Scores.
Acronym: Pawamedics
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Yorkshire Ambulance Service NHS Trust (Other Government)
Collaborators: National Institute for Health Research, United Kingdom (Other Government)
Responsible Party: Sponsor
Other Study IDs: YASRD170
Record Dates: First submitted 2022-06-24; First posted 2022-06-30 (Actual); Last update posted 2022-06-30 (Actual); Status verified 2022-06

CONDITIONS: Burn Out; EMS Exposures or Injuries of EMS Personnel
MeSH Terms: conditions — Burnout, Psychological

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Experimental Group: Ambulance Service Staff participating in pet therapy sessions.
  Interventions: Other: Copenhagen Burnout Inventry

INTERVENTIONS:
Other: Copenhagen Burnout Inventry — Questionnaire

SUMMARY:
Problem During the COVID 19 pandemic, NHS staff have become increasingly burned out. Mental health is the leading cause of staff sickness and absence in the NHS. Ambulance trusts have the highest rates of sickness across all NHS professions. Reduced staffing levels directly impacts service delivery. Staff struggling with poor mental health are more likely to make errors, have reduced empathy, and patients have lower patient satisfaction.

The Solution? Dog therapy is used in hospital settings around the world for patient benefit and staff welfare.

Evidence suggests dog therapy improves mood and reduces anxiety. Yorkshire Ambulance Service (YAS) has a small, but established dog therapy scheme, organised by the health and wellbeing team.

This research aims to observe if dog therapy affects symptoms of burnout in YAS staff. We will use two sets of staff:

Patient facing staff Staff with remote patient contact

What will participants need to do?

Participants will be given a Copenhagen Burnout Inventory - a questionnaire focusing on three factors:

Personal burnout Work related burnout Client related burnout

Burnout will be measured in 4 categories; no/low, moderate, high and severe burnout.

The questionnaire will be completed at the beginning and end of 8 weeks of dog therapy.

* Some optional demographic questions
* Number of sessions attended
* Engagement with occupational health services
* Dog Ownership

We will calculate the difference in severity of burnout between baseline and after 8 weeks of dog therapy.

A PPI group has been consulted on methodology, wording of plain English summary and the dissemination plan.

This research will be distributed to all interested participants, published in an appropriate journal presented at conferences, and presented in the ICA dissemination event.

ELIGIBILITY:
Inclusion Criteria:

Yorkshire Ambulance Service (YAS) Employee with patient contact. Patient contact includes face to face to face or remote patient contact. Taking part in YAS dog therapy scheme. Completed no more than 2 dog therapy sessions to date. -

Exclusion Criteria:

Staff with no patient contact as part of their role. Staff on bank contract

-

Ages: 18 Years to 68 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Convenience sample of patient facing staff who are participating in Yorkshire Ambulance Service pet therapy scheme.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2022-08-01 (Estimated); Primary Completion 2022-09-30 (Estimated); Study Completion 2022-09-30 (Estimated)

PRIMARY OUTCOMES:
Mean difference in change of each section of Copenhagen Burnout Inventory (CBI) Score | 8 weeks.
  CBI will be measured at week 0 and week 8. The CBI is composed of 3 sections. We will calculate a mean change in score for each of the 3 sections.

SECONDARY OUTCOMES:
Mean difference ambulance turnaround times. | 8 weeks.
  We will calculate a mean difference in ambulance turnaround times for those participating in dog therapy vs those not participating on dog therapy.
Drop out rate. | 8 weeks.
  We will report the proportion of participants that withdraw from the study.

CONTACTS AND LOCATIONS:
Overall Officials: Richard Pilbery, MSc, Principal Investigator — Yorkshire Ambulance Service NHS Trust

IPD SHARING:
Plan to Share IPD: Undecided